CLINICAL TRIAL: NCT00616824
Title: The Use of an Acellular Dermal Matrix in a Two-Staged Breast Reconstruction The Use of an Acellular Dermal Matrix in a Two-Staged Breast Reconstruction After Mastectomy: A Double-Blinded, Randomized Trial
Brief Title: The Use of an Acellular Dermal Matrix in a Two-Staged Breast Reconstruction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 070415; 070415
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Mastectomy; Postoperative Pain; Complications
Keywords: Acellular dermal matrix; breast reconstruction; tissue expander; postoperative pain; complication; pain; patient satisfaction
MeSH Terms: conditions — Pain, Postoperative; Pain; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional Method (Active Comparator): Arm which uses the Serratus Anterior muscle mobilization for lateral coverage of the tissue expander
  Interventions: Procedure: Serratus anterior to cover lateral aspect of tissue expander
- Dermamatrix Arm (Experimental): Arm which uses Dermamatrix as the lateral expander coverage
  Interventions: Procedure: Dermamatrix to cover lateral aspect of tissue expander

INTERVENTIONS:
Procedure: Dermamatrix to cover lateral aspect of tissue expander — Dermamatrix used to cover lateral aspect of breast tissue expander after mastectomy
  Other Names: Dermamatrix
  Arms: Dermamatrix Arm
Procedure: Serratus anterior to cover lateral aspect of tissue expander — Traditional use of serratus anterior for coverage of lateral aspect of tissue expander
  Arms: Traditional Method

SUMMARY:
This study intends to compare postoperative outcomes of a tissue expander placement following a mastectomy with two different operative techniques. This study will be randomized and double blinded comparing the traditional placement of the tissue expander under an inferolateral serratus muscle flap to a new technique which uses an acellular dermal matrix as an inferolateral sling, instead of the muscle flap.

The study we are proposing will evaluate the question of whether there is a difference between the traditional method of serratus flap and the new technique of using an acellular matrix with tissue expander placement. This will be a double blinded randomized study of thirty women in each group comparing outcomes which will include postoperative pain, complications (wound infection, hematoma, capsular contracture, etc), and patient satisfaction with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to Dr. Wendel's clinic who are older than 17 years of age undergoing a mastectomy and wish to have breast reconstruction with a tissue expander or those who have previously undergone a mastectomy and are now seeking reconstruction will be solicited for the study.

Exclusion Criteria:

* Preoperative radiation therapy
* Autoimmune disease
* Fever
* Uncontrolled diabetes mellitus
* Inability to comprehend or cooperate with postoperative instructions
* Local or systemic infection
* Have any allergies to the excipient ingredients found in the matrix
* Pregnancy
* Low vascularity of the surrounding tissue
* Mechanical trauma
* Poor nutrition
* Poor general medical condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
postoperative pain | perioperative up to 1 year

SECONDARY OUTCOMES:
aesthetic outcome | 1 year
complications (infection, hematoma, capsular contracture) | 1 year
Patient satisfaction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jason J. Wendel, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States